CLINICAL TRIAL: NCT01038518
Title: Health2010-14: Monitoring Biomarkers of Chronic Diseases in the General Population
Acronym: Health2010-4
Status: Completed | Type: Observational
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Steno Diabetes Centre, Gentofte, Denmark (Unknown)
Responsible Party: Principal Investigator, Allan Linneberg, Professor, Head of Section, Glostrup University Hospital, Copenhagen
Other Study IDs: H2009124
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Cardiovascular Disease; Type 2 Diabetes; Asthma; Allergy; Osteoporosis
Keywords: epidemiology; risk factors; micronutrients
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Asthma; Hypersensitivity; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Urine, serum, whole blood, extracted DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Health2010: Cross-sectional general population study

SUMMARY:
The overall aim of the Health2010-14 is to monitor the prevalence and trends of common chronic diseases (osteoporosis, diabetes, cardiovascular disease, asthma, allergy, and eczema) that are often un-diagnosed in the general population as well as biomarkers of micronutrient status. Specific aims include identification of novel lifestyle and genetic risk factors for the above diseases by investigating gene-lifestyle interactions.

DETAILED DESCRIPTION:
Over a 5-year period a series of population-based studies are carried out including a total of up to 10,000 persons aged 18-69 years selected from the general population of Copenhagen, Denmark. The study also include a follow-up of a previous population study (the Health2006). Participants complete questionnaires on health, lifestyle, and social factors and undergo a health examination including measurements of metabolic biomarkers, allergy tests, anthropometric measures, bioimpedance, biomarkers of micronutrients, spirometry.

ELIGIBILITY:
Inclusion Criteria:

* persons living in 10 municipalities of Copenhagen

Exclusion Criteria:

* pregnancy, non-Danish citizenship

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Random samples of persons living in 10 municipalities in the Western part of the Capital Region of Denmark (Copenhagen).
Sampling Method: Non-Probability Sample
Enrollment: 1522 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
5-year change in prevalence of biomarkers of chronic diseases (e.g. diabetes, asthma, allergy) and micronutrient status (e.g. vitamin D status). | 5 years

SECONDARY OUTCOMES:
significant interaction (on a additive scale) between Vitamin D status and genetic variants in the Vitamin D receptor in relation to selected chronic disease biomarkers | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Allan Linneberg, MD, PhD, Study Director — Research Center for Prevention and Health, Glostrup Hospital

REFERENCES:
- See also: Related Info — http://www.regionh.dk/fcfs